CLINICAL TRIAL: NCT00114647
Title: Procedures to Obtain Plasma, Lymphocytes, or Other Specimens for Research Studies
Brief Title: Apheresis to Obtain Plasma or White Blood Cells for Laboratory Studies
Status: Recruiting | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 810164; 81-I-0164
Record Dates: First submitted 2005-06-15; First posted 2005-06-16 (Estimated); Last update posted 2026-01-16 (Actual); Status verified 2025-08-21

CONDITIONS: Healthy Volunteers; HIV
Keywords: Blood Collection; Apheresis; Natural History

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1: Healthy Volunteers
- 2: HIV

SUMMARY:
This study will collect blood plasma and white blood cells from individuals using a procedure called apheresis. Apheresis is a method of collecting larger quantities of certain blood components that can safely be collected through a simple blood draw. The blood components will be used in laboratory research studies.

Patients 18 years of age and older who are currently enrolled in a NIH clinical research protocol may participate in this study. Relatives of patients and normal healthy volunteers will also be enrolled.

Individuals will undergo one of the following two apheresis procedures:

* Automated pheresis Blood is drawn through a needle placed in an arm vein and circulated through a cell separator machine. The plasma (liquid part of the blood) and white cells are extracted, and the red cells are re-infused into the donor through the same needle or a needle in the other arm. An anticoagulant (medication to prevent blood from clotting) is usually added to the blood while in the machine to prevent it from clotting during processing.
* Manual pheresis One unit (1 pint) of blood is drawn through a needle placed in an arm vein, similar to donating a pint of whole blood. The red blood cells, with or without plasma, are separated from the rest of the blood and returned to the donor through the same needle. Manual pheresis will be done only when a person s estimated total blood volume or red cell count is too low to safely permit removal of blood through a pheresis machine. An adult small in size or markedly anemic, for example, may fall into this category.

Some of the blood collected through apheresis may be stored for future studies of HIV disease and immune function and for HLA testing, a genetic test of markers of the immune system. Some of the blood may be used to screen for different types of viral liver infections, such as hepatitis A, B, C, D, E, F, or G.

...

DETAILED DESCRIPTION:
In order to carry out research procedures on the plasma or mononuclear components of blood, it is often necessary to obtain larger quantities of plasma or mononuclear cells than can be safely obtained by simple phlebotomy. These components can be easily and safely obtained using apheresis procedures in the Clinical Center Apheresis Unit. Other specimens are also sometimes needed for research, such as other blood components, body fluids (such as semen or urine) or secretions (from nose, mouth, or different skin areas). While this protocol is specifically designed to conform to the requirements of the Apheresis Unit for donors to have apheresis and other collection procedures, it also permits collection of these other donor specimens. However, the protocol, by itself, is not an independent research study but rather designed to facilitate sample collections that may aid other studies.

ELIGIBILITY:
* INCLUSION CRITERIA:

  18 years of age or older

Adequate venous access

Blood pressure less than or equal to 180/100; pulse rate 50-100, unless a lower pulse rate is considered normal for the volunteer (e.g. a conditioned athlete)

Adequate blood counts if undergoing apheresis (HIV positive volunteers and volunteers with vasculitis or other inflammatory diseases: hemoglobin greater than or equal to 9.0 g/dL, HCT greater than or equal to 28%, platelets greater than or equal to 50,000; HIV negative volunteers: hemoglobin greater than or equal to 12.5 g/dL, HCT greater than or equal to 38%, platelets greater than or equal to 150,000)

Willing and able to provide written informed consent, comply with study requirements and procedures, and comply with clinic policies (including stored samples, hepatitis screening, and genetic testing including HLA testing)

EXCLUSION CRITERIA:

Pregnant and/or breast-feeding women

Currently abusing alcohol or other drugs

Any medical condition for which the PI feels apheresis or other sample collection procedures might be contraindicated

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community Sample
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 1984-01-09 (Actual)

PRIMARY OUTCOMES:
Specimen collection for the study of infectious diseases | Ongoing
  Collection of specimens for the study of infectious diseases.

CONTACTS AND LOCATIONS:
Overall Officials: Susan L Moir, Ph.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Malaspina A, Moir S, Kottilil S, Hallahan CW, Ehler LA, Liu S, Planta MA, Chun TW, Fauci AS. Deleterious effect of HIV-1 plasma viremia on B cell costimulatory function. J Immunol. 2003 Jun 15;170(12):5965-72. doi: 10.4049/jimmunol.170.12.5965. PMID 12794123
- [Background] Moir S, Ogwaro KM, Malaspina A, Vasquez J, Donoghue ET, Hallahan CW, Liu S, Ehler LA, Planta MA, Kottilil S, Chun TW, Fauci AS. Perturbations in B cell responsiveness to CD4+ T cell help in HIV-infected individuals. Proc Natl Acad Sci U S A. 2003 May 13;100(10):6057-62. doi: 10.1073/pnas.0730819100. Epub 2003 May 1. PMID 12730375
- [Background] Migueles SA, Laborico AC, Shupert WL, Sabbaghian MS, Rabin R, Hallahan CW, Van Baarle D, Kostense S, Miedema F, McLaughlin M, Ehler L, Metcalf J, Liu S, Connors M. HIV-specific CD8+ T cell proliferation is coupled to perforin expression and is maintained in nonprogressors. Nat Immunol. 2002 Nov;3(11):1061-8. doi: 10.1038/ni845. Epub 2002 Oct 7. PMID 12368910
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_1981-I-0164.html